CLINICAL TRIAL: NCT06880224
Title: Intensive Combination Approach to Rollback the HIV Epidemic in Nigerian Youth (iCARE) Plus Effectiveness/Implementation Hybrid Study: Aim 2
Brief Title: Intensive Combination Approach to Rollback the HIV Epidemic in Nigerian Youth (iCARE) Plus Effectiveness/Implementation Hybrid Study
Acronym: iCARE Plus
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Northwestern University (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, Robert Garofalo, Professor, Northwestern University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: iCARE Plus; UG1HD113160 (NIH)
Record Dates: First submitted 2025-03-11; First posted 2025-03-17 (Actual); Last update posted 2025-03-17 (Actual); Status verified 2025-02

CONDITIONS: Adolescent HIV Infection
Keywords: Adolescents, HIV Testing, HIV Treatment

STUDY DESIGN:
Intervention Model Description: This is a hybrid effectiveness/implementation trial with an HIV Case Finding Intervention "Arm" and a parallel HIV Treatment Intervention "Arm" that is a randomized controlled trial.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- HIV Case Finding Intervention (Experimental): Combination HIV case finding and linkage to care intervention
  Interventions: Behavioral: Testing Peer navigation; Behavioral: PrEP Intervention; Behavioral: Social Media Outreach
- HIV Treatment Intervention (Experimental): Combination HIV treatment intervention vs. standard of care adherence among youth newly diagnosed with HIV and initiating ART
  Interventions: Behavioral: Treatment Peer Navigation; Behavioral: SMS Test messaging; Other: Adherence standard of care

INTERVENTIONS:
Behavioral: Testing Peer navigation — Peer navigators will promote HIV testing in YMSM and linkage to care if HIV-positive
  Arms: HIV Case Finding Intervention
Behavioral: PrEP Intervention — Motivational-interviewing to promote uptake of PrEP among those who test HIV-negative
  Arms: HIV Case Finding Intervention
Behavioral: Treatment Peer Navigation — Peer navigators will provide assistance and support to youth with HIV to optimize adherence to ART
  Arms: HIV Treatment Intervention
Behavioral: Social Media Outreach — Social media outreach to identify youth at risk for HIV
  Arms: HIV Case Finding Intervention
Behavioral: SMS Test messaging — Text (SMS) messages to remind and encourage youth to adhere to their ART
  Arms: HIV Treatment Intervention
Other: Adherence standard of care — Standard of care HIV treatment adherence
  Arms: HIV Treatment Intervention

SUMMARY:
Two combination interventions (HIV Case Finding Intervention and HIV Treatment Intervention), each with mHealth and Peer Navigation components, will be evaluated in two 48-week parallel hybrid effectiveness/implementation trials among youth aged 15-24 in Nigeria.

DETAILED DESCRIPTION:
Two combination interventions, each with mHealth and Peer Navigation components, will be evaluated in two 48-week parallel hybrid effectiveness/implementation trials among youth aged 15-24 in Nigeria:

1. HIV Case Finding Intervention: single arm trial of an HIV case finding and linkage to care intervention targeting young men at risk of HIV infection (n = 6000), particularly young men who have sex with men (YMSM) in Akwa Ibom, Benue, Enugu, Kano, Taraba, and Lagos states who complete HIV testing.

   Objectives: To determine the effectiveness of the intervention to:
   * identify youth living with HIV, particularly YMSM and
   * link those who test HIV-positive to HIV care
   * pre-exposure prophylaxis (PrEP) initiation (uptake) among those who test HIV-negative.
2. HIV Treatment Intervention: randomized controlled trial of a medication adherence and viral suppression intervention among youth newly diagnosed with HIV and initiating antiretroviral therapy (ART) for the first time (n = 600) at the participating clinical sites.

Objectives: To determine the effectiveness of the intervention on

* viral suppression and
* adherence to ART
* success of implementation in the target populations

ELIGIBILITY:
Inclusion Criteria:

HIV Case Finding Intervention:

* Aged 15 to 24
* Male birth sex of any current gender identity
* Understand basic English, Yoruba, Hausa, Igbo or Pidgin English For the PrEP component, must also be HIV-negative

HIV Treatment Intervention:

* Aged 15 to 24
* HIV seropositive
* Initiating ART for the first time at a Clinical Research Performance Site (CRPS) clinic or satellite clinic
* Understand basic English, Yoruba, Hausa, Igbo or Pidgin English
* Intention to remain a CRPS patient during follow-up

Exclusion Criteria:

* Unable to provide consent
* No parental permission if aged 15 and not emancipated

Ages: 15 Years to 24 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 500 (Estimated)
Dates: Start 2025-02-01 (Actual); Primary Completion 2028-08-31 (Estimated); Study Completion 2028-08-31 (Estimated)

PRIMARY OUTCOMES:
Case Finding: HIV-positive serostatus | 48 weeks
  HIV-positive serostatus based on rapid test with confirmation
Treatment: Viral suppression | 48 Weeks
  Viral suppression (< 200 copies per mL)

SECONDARY OUTCOMES:
Case Finding: Linkage to HIV care | 48 Weeks
  Linkage to HIV care within 30 days of positive HIV test
Case Finding: PrEP among youth who test HIV-negative | 48 weeks
  PrEP uptake among youth who test HIV-negative
Treatment: Adherence to antiretroviral therapy (ART) | 48 Weeks
  > 90% adherence to ART

CONTACTS AND LOCATIONS:
Overall Officials: Robert Garofalo, MD, Principal Investigator — Northwestern University
Locations (6):
- Nigeria (6):
  - University of Uyo Teaching Hospital, Uyo, Akwa Ibom State
  - Federal Medical Center, Makurdi, Benue State
  - University of Nigeria Teaching Hospital, Enugu, Enugu State
  - Aminu Kano Teaching Hospital, Kano, Kano State
  - Lagos University Teaching Hospital, Lagos, Lagos
  - Taraba State Specialist Hospital, Jalingo, Taraba State